CLINICAL TRIAL: NCT07334002
Title: A Randomized, Single-blind, Controlled Trial to Evaluate the Effects of Conventional Therapy on Tinnitus, Disability, and Quality of Life in Patients With Tinnitus
Brief Title: The Effects of Conventional Therapy on Tinnitus, Disability, and Quality of Life in Patients With Tinnitus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Roza Jizel Dagdelen MD, Medical Doctor , Assistant Researcher, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16.02.2021 / 3158
Record Dates: First submitted 2025-11-18; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-11

CONDITIONS: Tinnitus; Neural Therapy of Huneke
Keywords: Neural Therapy of Huneke; Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Anesthesia, Local; Betahistine; BID protein, human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental)
  Interventions: Procedure: Neural Therapy of Huneke
- Control Group (Active Comparator)
  Interventions: Drug: Betahistine 24 mg bid (Betaserc)

INTERVENTIONS:
Procedure: Neural Therapy of Huneke — The aim for tinnitus and facial pain is to regulate the trigeminal system and autonomic balance.
  Concentration used: Lidocaine 0.5%.
  The auriculotemporal, infraorbital, zygomaticotemporal, and stellate regions were targeted.
  Puncture applications: 0.3-0.5 mL will be administered behind the ear, around the mastoid process, behind the tragus, and in the temporomandibular region.
  If necessary, the stellate ganglion area can be supplemented with regulation injections.
  Negative aspiration and aseptic technique will be applied before each application.
  Transient mild dizziness or local redness may occur after application.
  To avoid the risk of systemic toxicity, the total dose should generally not exceed a maximum of 200 mg of lidocaine.
  Arms: Treatment Group
Drug: Betahistine 24 mg bid (Betaserc) — Patients will be given Betahistine 16-48 mg/day in divided doses, depending on their weight and disease severity.
  Arms: Control Group

SUMMARY:
A randomized, single-blind, controlled trial to evaluate the effects of neural therapy on tinnitus severity, disability, and quality of life in patients with tinnitus.

The study is planned to be conducted between December 2025 and March 2026. The sample size is 30 patients. The number of centers is 1. The study duration is 3 months.

DETAILED DESCRIPTION:
All patients with normal otologic examinations and a type A tympanogram will be included in the study. Those who meet the exclusion criteria will not be included in the study, and patients will be randomized. Subsequently, the groups will be divided into two groups: those who will receive only medical treatment and those who will receive neural therapy in addition to medical treatment. Patients will be administered tinnitus severity questionnaires based on the SF-12 (short form) and the VAS (visual analog scale), the Turkish adaptation of the Tinnitus Disability Inventory (THI). The same questionnaires will be administered at their follow-up visits three months later.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a type A tympanogram in the tympanogram of all cases with normal otological examinations (air-bone gap should not be observed in any case).

Exclusion Criteria:

* Patients with a disease that may cause objective tinnitus,

  * Otosclerosis,
  * Chronic otitis media,
  * Acoustic tumor,
  * Meniere's disease,
  * History of ear surgery or head trauma, and those with neuropsychiatric diseases.

Also:

* Patients who have had ear surgery,
* Permanent hearing loss (total),
* Severe cardiovascular system failure, uncontrolled arrhythmia,
* Severe renal failure, or liver failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Turkish version of the Tinnitus Disability Questionnaire (THI) | 3 months
SF-12 (short form) | 3 months
Tinnitus severity according to VAS (visual analog scale) | 3 months

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 6 months